CLINICAL TRIAL: NCT06784622
Title: Evaluatıon of the Effect of Pulpotomy Treatments Wıth Dıfferent Bıomaterıals on Postoperatıve Paın In Permanent Molars
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Fatma GURBUZ, research assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Pulpitis
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BİO MTA+ (CERKAMED, Poland) group (Experimental): Partial pulpotomy will be performed using bio mta+ (CERKAMED, Poland)
  Interventions: Drug: Treatment as usual
- Well-Root PT (Vericom Co., Chuncheon, Kore) group (Experimental): Partial pulpotomy will be performed using Well-Root PT
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Drug: Treatment as usual — Well-Root PT is clinically used in many areas such as pulp capping, perforation and resorption repair, root tip filling and apexification. As Well-Root PT is available in pre-mixed capsule form, it can provide a consistent and adequate consistency and clinical convenience. Well-Root PT can be applied directly into the oral cavity by placing the capsule in a syringe. In addition, Well-Root PT has a shorter setting time than MTA.Despite these advantages, there is no study in the literature on the effect of Well-Root PT on postoperative pain and tooth vitality after pulpotomy in mature permanent molars

SUMMARY:
The aim of this study was to evaluate the results of partial and total pulpotomy with mineral trioxide aggregate (BIO MTA+) and bioceramic sealer (Well Root PT) in terms of pain and vitality in permanent molars with exposed pulp due to caries.

DETAILED DESCRIPTION:
Dental caries, an infectious disease, is the most common cause of pulp inflammation. However, the dentin-pulp complex has several physiological defence mechanisms against caries. Preserving pulp viability is the primary goal of biologically based, minimally invasive treatments. Therefore, vital pulp treatments such as partial and total pulpotomies have become increasingly common. Vital pulp therapy is a series of conservative procedures that rely on the natural repair mechanisms of the dentin-pulp complex. This treatment is based on the placement of an appropriate medicamentous and sealed coronal restoration to create a biologically suitable environment for the pulp tissue to heal and protect against bacterial contamination. Root canal treatment is also commonly performed on teeth with deep caries. However, despite the high success rate of 89%, problems such as transpotation, apical zipper formation, instrument breakage during mechanical preparation, failure to reach all canals and inadequate or excessive root filling can lead to treatment failure. Unlike root canal treatment, which involves the removal of all pulp tissue, vital pulp treatment preserves the immune defence and regenerative potential of the pulp and allows root development to continue in immature teeth. Many studies show that the carious pulp of mature teeth is capable of regeneration and that vital pulp therapy is successful in symptomatic and permanent teeth . In recent years, calcium silicate-based cements (MTA, biodentin and bioceramic cements) have become the standard biomaterials for vital pulp treatment due to their biocompatibility and bioactivity . In vivo studies have shown predictable histological results in pulp healing with pulpotomy treatments using MTA . However, as MTA is manufactured in powder/liquid form, it requires a mixing procedure prior to application. As it is difficult to achieve the appropriate consistency of the powder/liquid ratio during the mixing process , changes in the mechanical or chemical properties of the materials may occur. A previous in vitro study found that changes in the powder/liquid ratio affected the radiopacity, setting time, solubility and calcium ion release of MTA. Well-Root PT (Vericom Co., Chuncheon, Korea), a premixed cement, has recently been introduced to the market. Well-Root PT is clinically used in many areas such as pulp capping, perforation and resorption repair, root tip filling and apexification. As Well-Root PT is available in pre-mixed capsule form, it can provide a consistent and adequate consistency and clinical convenience. Well-Root PT can be applied directly into the oral cavity by placing the capsule in a syringe. In addition, Well-Root PT has a shorter setting time than MTA (approximately 5 minutes for initial setting and 45 minutes for final setting) . Despite these advantages, there is no study in the literature on the effect of Well-Root PT on postoperative pain and tooth vitality after pulpotomy in mature permanent molars. Therefore, the aim of this study was to evaluate the effect of Well-Root PT on postoperative pain and tooth vitality in vivo in comparison with MTA (BIO MTA+).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with no significant health problems.
* Restorable and periodontally healthy teeth.
* Teeth with complete root development.
* Teeth with cold sensitivity and positive response to electric pulp testing.
* Lower jaw first and second molars with deep/extremely deep caries detected on periapical radiographs.

Exclusion Criteria:

* Patients with systemic diseases or allergic reactions
* Teeth with open apex
* Carious teeth that do not respond to pulp sensitivity tests
* Teeth without signs of bleeding after opening the pulp chamber.
* Detection of periodontal pockets with a depth greater than 4 mm.
* Teeth with suspected cracks or crown fractures.
* Severely damaged teeth
* Teeth whose bleeding cannot be controlledTeeth with open apex

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
assessment of postoperative pain with questionnaires | 12 month
  Visual Analogue Scala (VAS) will be used . 0: no pain 100: Worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry, Kayseri, melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No